CLINICAL TRIAL: NCT07393425
Title: Neoadjuvant Therapy With Trastuzumab Deruxtecan (SHR-A1811) + Pertuzumab or Trastuzumab Deruxtecan (SHR-A1811) + Pertuzumab Sequenced With Paclitaxel-based Regimens + Trastuzumab + Pyrotinib in HER2+ Breast Cancer
Brief Title: Neoadjuvant Trastuzumab Deruxtecan (SHR-A1811) + Pertuzumab in HER2+ Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kunwei Shen, Head of Comprehensive Breast Health Center, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBC2502
Record Dates: First submitted 2026-02-01; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: HER2 + Breast Cancer
Keywords: Trastuzumab Deruxtecan; SHR-A1811; neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; pertuzumab; Trastuzumab; Biosimilar Pharmaceuticals; pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Patients will receive three cycles of treatment with Trastuzumab Deruxtecan (SHR-A1811) + Pertuzumab, followed by imaging assessment. If clinical complete response (cCR) or radiological complete response/near radiological complete response (rCR/near rCR) is achieved, they will continue to receive an additional three cycles of treatment with Trastuzumab Deruxtecan (SHR-A1811) + Pertuzumab, followed by surgery.Patients who did not achieve cCR/rCR or near rCR at the end of cycle 3 will change to the THPy regimen (paclitaxel-based regimen + Trastuzumab + Pyrotinib) for three cycles.
  Interventions: Drug: Trastuzumab Deruxtecan; Drug: Pertuzumab; Drug: Taxane Chemotherapy; Drug: Trastuzumab (or biosimilar); Drug: Pyrotinib 320mg

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — 4.8mg/kg, d1, q3w
  Other Names: A1811
Drug: Pertuzumab — 840mg on cycle1, 420mg on following cycles, d1, q3w
Drug: Taxane Chemotherapy — Nab-paclitaxel 100 mg per square meter, d1,d8,d15 q3w Or Paclitaxel 80mg per square meter, d1,d8,d15 q3w Or Docetaxel 100mg per square meter, d1 q3w
Drug: Trastuzumab (or biosimilar) — Trastuzumab 8mg/kg (loading dose) or 6mg/kg on following cycles, d1, q3w
Drug: Pyrotinib 320mg — 320mg qd

SUMMARY:
Patients with Stage II-III HER2-positive breast cancer will receive three cycles of treatment with Trastuzumab Deruxtecan (SHR-A1811) + Pertuzumab, followed by imaging assessment. If clinical complete response (cCR) or radiological complete response/near radiological complete response (rCR/near rCR) is achieved, they will continue to receive an additional three cycles of treatment with Trastuzumab Deruxtecan (SHR-A1811) + Pertuzumab, followed by surgery.

If cCR/rCR or near rCR is not achieved, the treatment will be switched to the THPy regimen (paclitaxel-based regimen + Trastuzumab + Pyrotinib) for three cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age and Gender: Female patients aged ≥18 years and ≤70 years. Histological Confirmation: Patients must have histologically confirmed invasive breast cancer and must not have received any prior systemic anti-tumor therapy for breast cancer.
* HER2 Positivity: Histologically confirmed HER2 receptor positivity, following the 2018 ASCO-CAP HER2 positivity judgment guidelines.

Confirmed by pathology laboratory with immunohistochemistry (IHC) score of 3+, or 2+ with positive in situ hybridization (ISH) test (ISH amplification rate ≥2.0).

* Tumor Stage: Patients must have tumor staging conforming to the Stage II-III breast cancer criteria according to the eighth edition of the AJCC breast cancer TNM staging system (T1~T4, N1~N3, M0).
* Measurable Target Lesion: At least one measurable target lesion according to RECIST V1.1.
* ECOG Performance Status: ECOG functional status score of 0~1.
* Organ Function: Adequate organ function levels, with the following requirements (no blood transfusion or use of leukocyte or platelet elevation drugs within 2 weeks prior to screening):

  * Hematology: Absolute neutrophil count (ANC) > 1.5 × 109/L; Platelet count (PLT) > 75 × 109/L; Hemoglobin (Hb) > 90 g/L.
  * Blood Chemistry: Total bilirubin (TBIL) < 1.5 × ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 1.5 × ULN; Alkaline phosphatase < 2.5 × ULN; Blood urea nitrogen/urea (BUN/UREA) and creatinine (Cr) < 1.5 × ULN.
  * Cardiac Ultrasound: Left ventricular ejection fraction (LVEF) ≥ 55%.
  * 12-Lead ECG: Fridericia's method corrected QT interval (QTcF) < 470 msec.
* Reproductive Status: For premenopausal women with potential fertility, a pregnancy test must be performed within 7 days before treatment initiation, with negative serum/urine pregnancy results.
* Patients must not be lactating and must use adequate barrier contraception throughout the treatment cycle and for 6 months after treatment completion.

Voluntary Participation: Voluntary participation in the study with signed informed consent, good compliance, and willingness to cooperate with visit schedules and research-related procedures.

Exclusion Criteria:

* Stage IV Breast Cancer: Patients with Stage IV breast cancer. Inflammatory Breast Cancer: Patients with inflammatory breast cancer. Prior Malignancy Treatment: Patients who have received prior anti-tumor therapy or radiotherapy for any malignancy, or have concurrent other malignancies, excluding cured cervical intraepithelial neoplasia, basal cell carcinoma, or squamous cell carcinoma.
* Concurrent Anti-Tumor Therapy: Patients currently participating in other clinical trials involving anti-tumor therapy, including but not limited to chemotherapy, endocrine therapy, biological therapy, bone modification therapy, or immune checkpoint inhibitor therapy.
* Recent Surgery: Patients who have undergone major surgery unrelated to breast cancer within 4 weeks prior to the first dose of the study drug, or have not fully recovered from such surgery.
* Serious Cardiac Disease: Patients with serious cardiac conditions, including but not limited to:
* History of heart failure or systolic dysfunction (LVEF < 50%). Uncontrolled high-risk arrhythmia, such as atrial tachycardia, resting heart rate > 100 bpm, significant ventricular arrhythmia, or advanced atrioventricular block (i.e., Mobitz II second-degree or third-degree atrioventricular block).
* Angina pectoris requiring medication.
* Clinically significant heart valve disease.
* ECG showing transmural myocardial infarction.
* Uncontrolled hypertension (after medication, systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg).
* Uncontrolled Active Infection: Patients with uncontrolled active infection requiring treatment, or with a history of immunodeficiency, including HIV positivity, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
* Allergy to Study Drugs: Patients with a known history of allergy to any component of the study drugs.
* Pregnant or Lactating Women: Pregnant or lactating women, women of childbearing potential with positive baseline pregnancy test, or those unwilling to use effective contraception during the trial period and for 6 months after the last dose of the study drug.
* Interstitial Lung Disease: Patients with known or suspected interstitial lung disease; those with other severe pulmonary diseases that may interfere with drug-related pulmonary toxicity detection or management within 3 months prior to the first dose, including but not limited to idiopathic pulmonary fibrosis, organizing pneumonia/obliterative bronchiolitis, pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive/obstructive lung disease, or any pulmonary autoimmune or inflammatory disease such as rheumatoid arthritis, Sjögren's syndrome, or sarcoidosis; or those with a history of total pneumonectomy.
* Severe Concomitant Diseases: Patients with severe concomitant diseases or other conditions that may interfere with the planned treatment, or those deemed unsuitable for the study by the investigator for any other reason.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
pCR | after neoadjuvant treatment, at surgery
  ypT0/Tis ypN0

SECONDARY OUTCOMES:
ORR | after neoadjuvant treatment, at surgery
  ORR per RECIST v1.1
EFS | From enrollment to 5 years after surgery
  Event free survival
OS | From enrollment to 5 years after surgery
  Overall survival
bpCR | after neoadjuvant treatment, at surgery
  ypT0/is

OTHER OUTCOMES:
Incidence of Adverse events per NCI CTCAE 5.0 | From the day of first dose of study drug to 28 days after last dose of study drug, an average of 5 months
  Safety per NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine affiliated Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided